CLINICAL TRIAL: NCT00847795
Title: A Trial to Investigate the Accelerated Wound Healing and Antiscarring Potential, Safety, Toleration and Systemic Exposure of Intradermal RN1001 (Avotermin) in Male and Female Subjects Aged 60 Years and Over.
Brief Title: Efficacy and Safety of Intradermal RN1001 (Avotermin) in Elderly Subjects.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Renovo (Industry)
Responsible Party: Mark Cooper, Renovo Ltd
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: RN1001-319-1005
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Cicatrix
MeSH Terms: conditions — Cicatrix | interventions — TGFB3 protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): 5ng Avotermin
  Interventions: Drug: Avotermin
- 2 (Experimental): 50ng Avotermin
  Interventions: Drug: Avotermin
- 3 (Experimental): 100ng Avotermin
  Interventions: Drug: Avotermin
- 4 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 5 (No Intervention): Standard Care

INTERVENTIONS:
Drug: Avotermin — Intradermal administration
  Other Names: Juvista
  Arms: 1; 2; 3
Drug: Placebo — Placebo
  Arms: 4

SUMMARY:
An exploratory Phase-II trial with intradermal RN1001 (Avotermin) to investigate scar prevention and reduction and acceleration of healing. The trial has an additional objective to evaluate several different scar assessment techniques that can be used in future clinical trials in the prevention and reduction of scarring.

DETAILED DESCRIPTION:
Double blind, randomised, Placebo and Standard Care controlled, single centre study. Each subject receives a total of 6 wounds, two incisions and four punch biopsies. Each subject serves as their own control, i.e. Arm 1 incisions/biopsies randomly received one of two treatments and Arm 2 incisions/biopsies received the same treatments as for Arm 1 but in reverse. The randomisation of the treatment allowed for control of possible positional effects on healing/scarring. Healed scars from incisional wounds excised from Arm 1 and Arm 2 after 6 months for histological analysis.

ELIGIBILITY:
Inclusion Criteria:

* Clinically healthy, male and female subjects aged 60 years and over. All females will be at least 2 years post menopausal.
* Weight between 50 and 150kg or a body mass index within the permitted range for their height using Quetelet's index-weight (kg)/height²(m). The permitted index is between 15 - 35 kg/m2.

Exclusion Criteria:

* Subjects who on direct questioning and physical examination have a history or evidence of hypertrophic or keloid scarring or with tattoos or previous scars in the area to be biopsied.
* Subjects with a personal history of a bleeding disorder.
* Subjects with a skin disorder that is chronic or currently active and which the investigator considers will adversely affect the healing the acute wounds or involves the areas to be examined in this trial.
* Subjects with any clinically significant medical condition that would impair wound healing including renal, hepatic, haematological, neurological or immune disease.
* Subjects with a history of clinically significant drug hypersensitivity to lignocaine or allergy to surgical dressings to be used in this trial.
* Subjects with any clinically significant abnormality following review of pre trial laboratory data and physical examination (see above).
* Subjects who are taking, or have taken, any investigational drugs, long term oral, topical or inhaled corticosteroid therapy, hormone replacement therapy (HRT) or anti-coagulant drugs in the thirty days prior to Day 0.
* Subjects who have evidence of drug abuse.
* Subjects who are known to have or had serum hepatitis or who are carriers of the hepatitis B surface antigen or hepatitis C antibody. Subjects with previous vaccination against Hepatitis B are not excluded per se.
* Subjects who are known to have or had serum hepatitis or who are carriers of the hepatitis B core antibody and who show less than 10 units per litre of Anti-HBs.
* Subjects who have previously had a positive result to the test for HIV antibodies, or who admit to belonging to a high-risk group.
* In the opinion of the investigator, a subject who is not likely to complete the trial for what ever reason.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2002-09; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of scar appearance by an independent panel | 6 months

SECONDARY OUTCOMES:
Histological evaluation of wound healing | 3 days
Adverse event occurance | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Duncan, BS BCh, Principal Investigator — Renovo
Locations (1):
- Renovo CTU, Manchester, United Kingdom

REFERENCES:
- [Derived] Ferguson MW, Duncan J, Bond J, Bush J, Durani P, So K, Taylor L, Chantrey J, Mason T, James G, Laverty H, Occleston NL, Sattar A, Ludlow A, O'Kane S. Prophylactic administration of avotermin for improvement of skin scarring: three double-blind, placebo-controlled, phase I/II studies. Lancet. 2009 Apr 11;373(9671):1264-74. doi: 10.1016/S0140-6736(09)60322-6. PMID 19362676